CLINICAL TRIAL: NCT04510571
Title: Evaluation of Postoperative Pain and Instrumentation Time After Root Canal Treatment With Rotary and Reciprocal File Systems in Children - A Randomized Clinical Trial
Brief Title: Evaluation of Postoperative Pain in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Alp Abidin Ateşçi, Principal Investigator, Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 20-7T/55
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Postoperative Pain
Keywords: postoperative pain; root canal treatment; reciprocal motion; rotary motion
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protaper Next (Active Comparator): Protaper Next group (n=25): The instrumentation of mesial and distal canals were done according to manufacturer's recommendations using X1 and X2 (25.06) at a rotational speed of 300 rpm. Then X3 and X4 (40.06) instruments were used to enlarge distal canals in order to compare the results with the Reciproc Blue group. The root canals were irrigated with 2 ml of %2,5 sodium hypochlorite after each instrument exchange.
  Interventions: Other: Evaluating Postoperative Pain After Root Canal Treatment with Protaper Next
- Reciproc Blue (Active Comparator): Reciproc Blue group (n=25) : The canals were shaped with in accordance with the manufacturer's recommendations. R25 (25.08) instrument was introduced into the canal with slow pecking movement within a 3 mm range each time. The flutes and remnants were cleaned after 3 pecking moves. Then R40 instrument (40.06) was selected to shape the distal canals as the #20 K file was passively introduced to the working length. The root canals were irrigated with 2 ml of %2,5 sodium hypochlorite after each instrument exchange.
  Interventions: Other: Evaluating Postoperative Pain After Root Canal Treatment with Reciproc Blue Files

INTERVENTIONS:
Other: Evaluating Postoperative Pain After Root Canal Treatment with Protaper Next — Patients were randomly separated into two groups and root canal treatments were completed with Protaper Next file systems. Instrumentation time for each system was noted and patients were given a pain scale which included visual analog scale for 6, 24, 48 and 72 hours after treatment.Postoperative pain scores and instrumentation times were analyzed statistically with chi square test and student t test.
  Other Names: Root Canal Instrumentation; Root Canal Treatment; Assessing Postoperative Pain; Instrumentation Time
  Arms: Protaper Next
Other: Evaluating Postoperative Pain After Root Canal Treatment with Reciproc Blue Files — Patients were randomly separated into two groups and root canal treatments were completed with Reciproc Blue file systems. Instrumentation time for each system was noted and patients were given a pain scale which included visual analog scale for 6, 24, 48 and 72 hours after treatment.Postoperative pain scores and instrumentation times were analyzed statistically with chi square test and student t test.
  Other Names: Root Canal Instrumentation; Root Canal Treatment; Assessing Postoperative Pain; Instrumentation Time
  Arms: Reciproc Blue

SUMMARY:
Postoperative pain is a common symptom of a flare up after root canal treatments (RCTs). Insufficient instrumentation, extrusion of irrigation solutions and debris and existence of a periapical lesion are the factors affecting postoperative pain after root canal treatments. Aim of this study is to evaluate the postoperative pain and instrumentation time of single-file reciprocating system and multiple-file Ni-Ti rotary system in children ages between 9-12. Study was conducted on fifty first permanent mandibular molars with the diagnosis of irreversible pulpitis. Patients were randomly separated into two groups and RCTs were completed with either Reciproc Blue or Protaper Next file systems. Instrumentation time for each system was noted and patients were given a pain scale which included visual analog scale for 6, 24, 48 and 72 hours after treatment. Postoperative pain scores and instrumentation times were analyzed statistically with chi square test and student t test. There was no statistically significant difference in postoperative pain between Reciproc Blue and Protaper Next systems at all time intervals. Instrumentation time was significantly shorter in the Reciproc Blue group in comparison with the Protaper Next group. In conclusion, shorter treatment time of single-file reciprocating systems may be more patient friendly and comfortable than multiple-file rotary systems in RCTs among children.

ELIGIBILITY:
Inclusion Criteria:

* Patients with first permanent mandibular molar teeth which had been diagnosed with symptomatic irreversible pulpitis with no periapical pathology or abscess were included in the study.

Exclusion Criteria:

* Patients who were on antibiotics or analgesics preoperatively were not included in the study.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Assessment After 6 hours | 6 hours after treatment
  Postoperative pain scores were scored using Modified Wong Baker pain rating scale (0 = no pain, 1 = slight pain, 2 = moderate pain, 3 = severe pain).
Postoperative Pain Assessment After 24 hours | 24 hours after treatment
  Postoperative pain scores were scored using Modified Wong Baker pain rating scale (0 = no pain, 1 = slight pain, 2 = moderate pain, 3 = severe pain).
Postoperative Pain Assessment After 48 hours | 48 hours after treatment
  Postoperative pain scores were scored using Modified Wong Baker pain rating scale (0 = no pain, 1 = slight pain, 2 = moderate pain, 3 = severe pain).
Postoperative Pain Assessment After 72 hours | 72 hours after treatment
  Postoperative pain scores were scored using Modified Wong Baker pain rating scale (0 = no pain, 1 = slight pain, 2 = moderate pain, 3 = severe pain).

SECONDARY OUTCOMES:
Instrumentation Time | During procedure
  The time for root canal instrumentation was recorded after working length determination until the end of instrumentation including irrigation between file changes within the sequence.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sathorn C, Parashos P, Messer H. The prevalence of postoperative pain and flare-up in single- and multiple-visit endodontic treatment: a systematic review. Int Endod J. 2008 Feb;41(2):91-9. doi: 10.1111/j.1365-2591.2007.01316.x. Epub 2007 Oct 23. PMID 17956561
- [Result] Cicek E, Kocak MM, Kocak S, Saglam BC, Turker SA. Postoperative pain intensity after using different instrumentation techniques: a randomized clinical study. J Appl Oral Sci. 2017 Jan-Feb;25(1):20-26. doi: 10.1590/1678-77572016-0138. PMID 28198972
- [Result] Shokraneh A, Ajami M, Farhadi N, Hosseini M, Rohani B. Postoperative endodontic pain of three different instrumentation techniques in asymptomatic necrotic mandibular molars with periapical lesion: a prospective, randomized, double-blind clinical trial. Clin Oral Investig. 2017 Jan;21(1):413-418. doi: 10.1007/s00784-016-1807-2. Epub 2016 Apr 4. PMID 27041109